CLINICAL TRIAL: NCT00005923
Title: The Effect of Estrogen and Progesterone Levels on Knee and Ankle Joint Laxity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00109-0749; M01RR000109 (NIH)
Record Dates: First submitted 2000-06-23; First posted 2000-06-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Healthy
Keywords: Joint Instability
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
The proposed research is an observational study designed to compare estrogen and progesterone serum levels with knee and ankle joint laxity, and muscle reaction time as a measure of neuromuscular function. Three groups of women athletes with differing estrogen and progesterone profiles (normal menstrual cycles, amenorrheic, and exogenous estrogen supplementation) and one control group (male collegiate athletes) will be used to compare differences in joint laxity and neuromuscular function. Blood levels of estrogen and progesterone will be measured at four time points across the menstrual cycle. Joint laxity and muscle reaction time will also be measured at each of these points. The investigator hypothesizes that knee and ankle joint laxity and muscle reaction time will significantly increase with increasing estrogen and progesterone levels.

ELIGIBILITY:
Inclusion Criteria:

* pre-collegiate or collegiate athletes

Ages: 15 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States